CLINICAL TRIAL: NCT04190316
Title: Study of the Fecal Relative Abundance (RA) of ESBL-producing Enterobacteriaceae (ESBL-PE) in Intensive Care (BLSE-REA) : What Are the Factors Influencing the Fecal RA of ESBL-PE in ICU ?
Brief Title: Factors Influencing the Fecal Relative Abundance of ESBL-producing Enterobacteriaceae in Intensive Care (BLSE-REA).
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RCB 2019-A02861-56
Record Dates: First submitted 2019-12-02; First posted 2019-12-09 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: ESBL-producing Enterobacteriaceae Infections
Keywords: Extended-spectrum beta-lactamase; Carriage; Cross transmission; Intensive care unit; Fecal relative abundance
MeSH Terms: interventions — Intensive Care Units

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluation of patient and patient-care environment ESBL (Other): ESBL-PE carriers included in the study will be sampled for evaluation of their fecal RA of ESBL-PE on day 0, 3, 5, 7, 10, 14 and weekly till day 30 or their discharge from ICU. Urine and respiratory samples will be collected on the same day to identify multiple-site colonization with ESBL-PE. Seven samples of patient care environment will be performed 2-times a week till day 30 or discharge of the patient from the ICU.
  Interventions: Other: Evaluation of fecal RA and environmental contamination of ESBL-PE carrier in ICU

INTERVENTIONS:
Other: Evaluation of fecal RA and environmental contamination of ESBL-PE carrier in ICU — ESBL-PE carriers included in the study will be sampled for evaluation of their fecal RA of ESBL-PE on day 0, 3, 5, 7, 10, 14 and weekly till day 30 or their discharge from ICU. Urine and respiratory samples will be collected on the same day to identify multiple-site colonization with ESBL-PE. Seven samples of patient care environment will be performed 2-times a week till day 30 or discharge of the patient from the ICU.

SUMMARY:
Extended-Spectrum Beta-Lactamases (ESBL)-Producing Enterobacteriaceae (PE) pose a major problem among antimicrobial resistance. The worldwide spread of theses bacteria may be responsible for 10 million death in 2050. Infection with ESBL-PE are associated with a worse prognosis because of delay in the start of adequate antibiotic treatment, especially for severe infections. It has been proposed to identify colonized patients to predict the risk of infection and the risk of nosocomial cross transmission.

This qualitative approach has limit as only 5 to 20% of patients will develop an infection with ESBL-PE. The fecal relative abundance (RA) of ESBL-PE is a ratio of ESBL-PE among enterobacteriaceae that could identify high-risk patients of infection or cross transmission. ESBL-PE RA may be highly variable in patient with antibiotic exposure depending on the molecule received but dynamic data is missing.

The aim of this study is to identify the factor that influence the fecal RA of ESBL-PE in ICU and to evaluate the association between different level of fecal RA and infection or cross transmission with an ESBL-PE.

DETAILED DESCRIPTION:
Antimicrobial resistance is rising since decades with a risk of million of death in the future. Extended-Spectrum Beta-Lactamases (ESBL)-Producing Enterobacteriaceae (PE) have expanded exponentially since 15 years and represent with Carbapenemase-PE one of the major challenges in resistance control. The burden of ESBL-PE infections is major in intensive care units (ICU) because of the delay to identify an effective antibiotic treatment (highly associated with outcome) and because of a higher risk of nosocomial cross transmission.

Identification of digestive carrier of ESBL-PE is based on a qualitative result that categorize the patient as a carrier or as non-carrier. This result makes it impossible to individualize the measures to be taken for an ESBL-PE carrier.

Prevention of cross transmission has no formal guideline. Some practitioners in ICU have stopped to detect for ESBL-PE carriage (specially when prevalence is low) and other prefer to close the ward (specially during outbreak).

Empiric treatment of most infections in ESBL-PE carrier are based on last-resort antibiotic (i.e. carbapenem) until microbiological results of a clinical simple is available.

A quantitative approach based on fecal relative abundance (RA) of ESBL-PE (ratio between ESBL-PE and enterobacteriaceae) has been proposed to individualize the risk of urinary tract infection (UTI) for ambulatory patients. In this setting, a fecal carriage with a very low RA of ESBL-PE safely rule out a risk of infection with ESBL-PE and patients with a high RA had an increased risk of UTI infection with ESBL-PE. Large variations of RA ESBL-PE carriage was observed and prediction of the level of RA was not possible for a patient.

A high variation in fecal RA of ESBL-PE is probable in ICU because of a high proportion of antibiotic exposure. Using the RA in ICU for ESBL-PE carrier could make it possible to identify patients who need for carbapenem in their empiric treatment and those who need continuing contact precautions to prevent cross transmission.

The aim of this study is to identify the factor that influence the fecal RA of ESBL-PE in ICU and to evaluate the association between different level of fecal RA and infection or cross transmission with an ESBL-PE.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Positive sample for ESBL-PE at admission of during ICU stay
* Patient's or relative's consent

Exclusion Criteria:

* Women pregnant, parturient or breast-feeding during the study period
* Patient deprived of liberty by judicial or administrative decision
* Patient undergoing psychiatric care under duress
* Patient subject to a legal protection measure
* Patient with no social security coverage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Changes in fecal ESBL-PE RA in the ICU | Day 0, 3, 5, 7, 10, 14 and weekly till day 30.
  Factors associated with changes in the RA of ESBL-PE fecal carriage will be analyzed. RA is expressed by the ratio of ESBL-PE and total enterobacteriaceae.

SECONDARY OUTCOMES:
Association between changes in ESBL-PE RA in fecal samples and ESBL-PE infection | Day 0, 3, 5, 7, 10, 14 and weekly till day 30.
  Looking for a threshold of ESBL-PE RA in fecal sample and a high risk of ESBL-PE infection
Association between changes in ESBL-PE RA in fecal samples and ESBL-PE cross-transmission | Day 0, 3, 5, 7, 10, 14 and weekly till day 30.
  Is there an association between a high ESBL-PE RA in fecal samples and cross-transmission
Association between changes in ESBL-PE RA in fecal samples and multiple-site colonization | Day 0, 3, 5, 7, 10, 14 and weekly till day 30.
  Is there an association between a high ESBL-PE RA in fecal samples and multiple-site colonization
Association between changes in ESBL-PE RA in fecal samples and patient care environment contamination with ESBL-PE | Twice a week till day 30.
  Is there an association between a high ESBL-PE RA in fecal samples and patient care environment contamination with ESBL-PE
Comparison of changes in ESBL-PE RA between different bacteria species during ICU stay | Day 0, 3, 5, 7, 10, 14 and weekly till day 30.
  Are there differences of RA between different species of ESBL-PE
Incidence of high level of EBSL-PE RA in ICU fecal carriers | Day 0, 3, 5, 7, 10, 14 and weekly till day 30.
  High level of RA is defined by a ratio of ESBL-PE on total enterobacteriaceae > 0.2

IPD SHARING:
Plan to Share IPD: No